CLINICAL TRIAL: NCT02411383
Title: Prospective, Single-centre, Open-label Clinical Study to Investigate the Safety and Performance of the NeuRx Diaphragm Pacing System (DPS) in Patients Undergoing Bilateral Lung Transplantation
Brief Title: Clinical Study to Investigate Safety and Performance of NeuRx DPS in Patients Undergoing Bilateral Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-1000-0001
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: Diaphragm pacing; Respiratory assistance; Lung transplant
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeuRx Diaphragm Pacing System (DPS)® (Experimental): The NeuRx Diaphragm Pacing System (DPS)® is placed in the diaphragm during lung transplant.
  Interventions: Device: NeuRx Diaphragm Pacing System

INTERVENTIONS:
Device: NeuRx Diaphragm Pacing System — NeuRx Diaphragm Pacing System electrodes are placed in the diaphragm during lung transplant surgery. The diaphragm will be continually paced until the patient is free from the ventilator or the patient is discharged from the ICU whichever. Diaphragm measurements are taken daily to assess tolerability and pacing success.

SUMMARY:
This study is a prospective, single-center feasibility study to acquire more knowledge regarding the NeuRx DPS and develop a routine in the optimal pacing of the diaphragm with this system during the weaning period from mechanical ventilation in the Intensive Care Unit in patients after bilateral lung transplant.

DETAILED DESCRIPTION:
This study is a prospective, single-center feasibility study to acquire more knowledge regarding the NeuRx DPS and develop a routine in the optimal pacing of the diaphragm with this system during the weaning period from mechanical ventilation in the Intensive Care Unit in patients after bilateral lung transplant. The objectives are to evaluate the safety and technical performance of DPS by assessing:

* the immediate safety and technical surgical results of implantation
* the safety and tolerability of use and removal until patient discharge from the Intensive Care Unit (ICU) or hospital
* the effects of diaphragm pacing on MV interaction, diaphragm force, fatigue resistance, and diaphragm electromyography (EMG)

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing bilateral lung transplantation
* Signed written informed consent has been obtained prior to any study related procedure

Exclusion Criteria:

* Diaphragm malformation which makes the electrode insertion impossible
* Presence of contra-indications for magnetical stimulation; pacemaker or implantable cardioverter-defibrillator, prosthetic valve, cervical implants, cervical trauma
* Participation in other clinical studies that could interfere with the results in the ongoing study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety: Daily assessment of device or procedure-related adverse events until patient discharge. | 30 days
Tolerability: Patient withdrawal from treatment. | 30 days
Pacing success: Ability to ventilate the patient through diaphragm pacing with or without assistance of mechanical ventilation. | 30 days

SECONDARY OUTCOMES:
Composite endpoint | 30 days
  Effects of diaphragm pacing on MV interaction, diaphragm force, fatigue resistance, and diaphragm electromyography (EMG).

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium